CLINICAL TRIAL: NCT00327340
Title: Title: A Pilot Study Evaluating the Safety and Feasibility of Custirsen (OGX-011) in Combination With Second Line Chemotherapy in Patients With Hormone Refractory Prostate Cancer
Brief Title: Evaluation of Safety and Feasibility of OGX-011 in Combination With 2nd-line Chemotherapy in Patients With HRPC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Achieve Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OGX-011-07
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: Metastatic hormone refractory prostate cancer (HRPC)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — OGX-011

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OGX-011 / mitoxantrone/prednisone (Experimental): OGX-011 / mitoxantrone/prednisone: OGX-011 administered in combination with mitoxantrone and prednisone
  Interventions: Drug: custirsen (OGX-011)/mitoxantrone
- OGX-011/docetaxel/prednisone (Experimental): OGX-011/docetaxel/prednisone: OGX-011 administered in combination with docetaxel and prednisone
  Interventions: Drug: custirsen (OGX-011)/docetaxel

INTERVENTIONS:
Drug: custirsen (OGX-011)/mitoxantrone — All subjects began treatment with oral prednisone (5 mg twice daily, 10 mg/day) continued through completion of the final treatment cycle. Three IV administrations of OGX-011 (640 mg) were given as 2 hr infusions during the loading dose period (Days-9 to-1). Subjects were premedicated with either ibuprofen (400 mg) or acetaminophen (650 mg) 30 to 60 minutes prior to and every 4-6 hours for 24 hours following each of the three doses of OGX-011 during the loading dose period only. After the loading dose period, OGX-011 was given weekly on Days 1, 8, and 15 of each 21-day cycle.
  Mitoxantrone was administered IV on Day 1 of each cycle at a planned dose of 12 mg/m² infused over 30 minutes.
  Patients could receive a maximum of 9 cycles of treatment.
  Other Names: custirsen; OGX-011; TV-1011
  Arms: OGX-011 / mitoxantrone/prednisone
Drug: custirsen (OGX-011)/docetaxel — All subjects began treatment with oral prednisone (5 mg twice daily, 10 mg/day) continued through completion of the final treatment cycle. Three IV administrations of OGX-011 (640 mg) were given as 2 hr infusions during the loading dose period (Days-9 to -1). Subjects were premedicated with either ibuprofen (400 mg) or acetaminophen (650 mg) 30 to 60 minutes prior to and every 4-6 hours for 24 hours following each of the three doses of OGX-011 during the loading dose period only. After the loading dose period, OGX-011 was given weekly on Days 1, 8, and 15 of each 21 day cycle.
  Docetaxel was administered IV on Day 1 of each cycle at a planned dose of 75 mg/m² infused over 60 minutes.
  Patients could receive a maximum of 9 cycles of treatment.
  Other Names: custirsen; OGX-011; TV-1011
  Arms: OGX-011/docetaxel/prednisone

SUMMARY:
This study is for patients with cancer of the prostate gland that has metastasized or spread outside the prostate to other parts of the body. Patients have already been treated with a drug called docetaxel or Taxotere® (with or without the addition of a steroid called prednisone) some time in the recent past. They either did not respond to this therapy or responded to this therapy, but now the cancer is progressing (growing larger or has spread to other areas of the body).

Custirsen (OGX-011) is an experimental drug that has been shown to increase the effectiveness of chemotherapy in several kinds of tumors, including prostate cancer.

Both docetaxel and mitoxantrone have anticancer activity in prostate and are approved by Health Canada and the Food and Drug Administration for the treatment of patients with prostate cancer.

DETAILED DESCRIPTION:
This study was initiated as a multicenter, open-label, randomized study, with a planned enrollment of 40 subjects. Although two treatment arms were included in this study, no comparison between the arms was intended.

Subjects with metastatic HRPC who failed first-line docetaxel therapy and required second-line therapy were randomly assigned to treatment with OGX-011 in combination with docetaxel/prednisone (OGX-011/docetaxel/prednisone) or OGX-011 in combination with mitoxantrone/prednisone (OGX-011/mitoxantrone/ prednisone). The study was randomized to assure that subjects were enrolled in each of the two treatment arms in an unbiased manner.

Based on preliminary safety data from the first 44 subjects who were randomized to receive either docetaxel or mitoxantrone, the protocol was amended to enroll approximately 20 additional subjects who would be assigned to the docetaxel/prednisone treatment arm to further investigate safety of the combination.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologic diagnosis of adenocarcinoma of the prostate.
3. Metastatic disease on chest X-ray, bone scan, or computed tomography (CT) scan.
4. Failed after receiving a minimum of two cycles of a docetaxel based first line therapy regimen. Failure is defined as disease progression within 6 months of discontinuing first line docetaxel therapy. Disease progression is defined as one or more of the following:

   * Progressive measurable (target) disease (by Response Evaluation Criteria in Solid Tumors [RECIST] criteria): at least a 20% increase in the sum of the longest diameters of measurable lesions (organ masses or lymph nodes) over the smallest sum observed (baseline or nadir) or the appearance of one or more new lesions as assessed by CT scan or chest X-ray.
   * Bone scan progression: one or more new lesions on bone scan while on or following docetaxel treatment.
   * Increasing serum PSA level: rise in PSA on three consecutive measurements obtained at least one week apart. If the third PSA value is less than the second, an additional fourth test to confirm a rising PSA will be acceptable.
5. Baseline laboratory values as stated below:

   * Creatinine ≤ 1.5 x upper limit of normal (ULN)
   * Bilirubin ≤ 1.1 x ULN (unless elevated secondary to conditions such as Gilbert's disease)
   * SGOT (AST) ≤ 1.5 x ULN
   * Castrate serum testosterone level (< 50 ng/mL-or-< 1.7 mmol/L).
6. If not treated with bilateral orchiectomy, patients must be willing to continue luteinizing hormone releasing hormone analogues throughout the study.
7. Adequate bone marrow function defined as absolute neutrophil count (ANC) ≥ 1.5 x 10^9 cells/L and platelet count ≥ 100 x 10^9/L.
8. Karnofsky score ≥ 60
9. Received no other chemotherapy, radioisotope therapy, strontium 89, or samarium 153. (Prior radiotherapy and steroids following first line docetaxel therapy are allowed.)
10. Received no more than one prior biological response modifier therapy following first line docetaxel therapy.
11. At least 21 days since completing the last dose of docetaxel, biological response modifier, and/or radiotherapy. (Exception for radiotherapy: at least 7 days since completing a single fraction of ≤ 800 cGy to a restricted field.)
12. Has recovered from all therapy related toxicity to ≤ grade 2, (except alopecia and anemia.)
13. Willing and able to give informed consent and follow protocol requirements.

Exclusion Criteria:

1. Life expectancy less than 12 weeks.
2. Patient is beyond 6 months following the last dose of docetaxel.
3. Patient could not tolerate a dose of docetaxel of at least 45 mg/m² at the end of first line therapy due to toxicity.
4. History of or current documented brain metastasis or carcinomatous meningitis, treated or untreated. (Brain imaging in asymptomatic patients is not required.)
5. Current symptomatic cord compression requiring surgery or radiation therapy. (Once treated, patients are eligible for the study.)
6. Active second malignancy (except non melanomatous skin or superficial bladder cancer).
7. Prior radiotherapy to > 25% of the bone marrow.
8. Uncontrolled medical conditions such as a major active infection, myocardial infarction or stroke within 3 months, uncontrolled hypertension, and/or significant concurrent medical illness, that, in the opinion of the Investigator, would preclude protocol therapy.
9. History of or active congestive heart failure.
10. Known allergy or hypersensitivity to docetaxel or polysorbate 80 (diluent).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Saad, MD, FRCS, Principal Investigator — Université de Montréal; Eric Winquist, MD, MSc, Principal Investigator — Western University, Canada
Locations (10):
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Toronto Sunnybrook, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - University of Montreal, Montreal, Quebec

REFERENCES:
- [Result] Saad F, Hotte S, North S, Eigl B, Chi K, Czaykowski P, Wood L, Pollak M, Berry S, Lattouf JB, Mukherjee SD, Gleave M, Winquist E; Canadian Uro-Oncology Group. Randomized phase II trial of Custirsen (OGX-011) in combination with docetaxel or mitoxantrone as second-line therapy in patients with metastatic castrate-resistant prostate cancer progressing after first-line docetaxel: CUOG trial P-06c. Clin Cancer Res. 2011 Sep 1;17(17):5765-73. doi: 10.1158/1078-0432.CCR-11-0859. Epub 2011 Jul 25. PMID 21788353
- [Derived] Blumenstein B, Saad F, Hotte S, Chi KN, Eigl B, Gleave M, Jacobs C. Reduction in serum clusterin is a potential therapeutic biomarker in patients with castration-resistant prostate cancer treated with custirsen. Cancer Med. 2013 Aug;2(4):468-77. doi: 10.1002/cam4.93. Epub 2013 May 28. PMID 24156019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 10 institutions with a primary focus in oncology and located in Canada. The first subject was randomized on July 25, 2006. The last subject completed treatment on August 6, 2008 and the last survival follow-up visit was on August 13, 2010
Pre-assignment Details: A total of 70 subjects were enrolled. 45 subjects were randomly assigned to treatment (21 to OGX-011/ docetaxel and 24 OGX-011/ mitoxantrone). An additional 25 subjects were enrolled under Amendment 2 and assigned to OGX-011/docetaxel retreatment. One subject was found to be ineligible and was not treated.
Groups:
- OGX-011 / Mitoxantrone/Prednisone: All subjects began with oral prednisone (5 mg twice daily)on Day-10. Custirsen (OGX-011) was infused intravenously over 2 hours on Day -7, -5 and-3 of cycle 1 (Pretreatment loading doses). OGX-011 was then infused for 2 hours on Days 1, 8, and 15 of each 21-day cycle. Mitoxantrone was infused at a dose of 12 mg/m² over 30 minutes on day 1 of each cycle.
- OGX-011 / Docetaxel/Prednisone: All subjects began with oral prednisone (5 mg twice daily)on Day-10. Custirsen (OGX-011) was infused intravenously over 2 hours on Day -7, -5 and -3 of cycle 1 (Pretreatment loading doses). OGX-011 was then to be infused for 2 hours on Days 1, 8, and 15 of each 21-day cycle. Docetaxel was infused at a dose of 75 mg/m² over 60 minutes on day 1 of each cycle.
Period: Overall Study
Arm/Group | OGX-011 / Mitoxantrone/Prednisone | OGX-011 / Docetaxel/Prednisone
Started | 23 | 46
Completed | 8 | 16
Not Completed | 15 | 30
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Physician Decision | 1 | 1
Not completed — Disease Progression | 10 | 19
Not completed — Symptomatic Disease | 0 | 2
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OGX-011 / Mitoxantrone/Prednisone | OGX-011 / Docetaxel/Prednisone | Total
Number analyzed (Participants) | 23 | 46 | 69
Age Continuous [Median (Full Range); unit: years] | 61 [49 to 81] | 64 [48 to 80] | 63 [48 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 23 | 46 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 21 | 42 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Karnofsky Score [Number; unit: participants] — The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment.
  100%=Normal no complaints; no evidence of disease 90%=Able to carry on normal activity; minor signs or symptoms of disease 80%=Normal activity with effort;some signs or symptoms of disease 60-70%=Able to care for self;unable to do active work
  participants
    60-70% | 2 | 6 | 8
    80% | 7 | 13 | 20
    90% | 7 | 22 | 29
    100% | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Custirsen (OGX-011) in Combination With Either Docetaxel/Prednisone or Mitoxantrone/Prednisone as Second-line Chemotherapy.
Description: Safety and tolerability were based on Adverse Events (AE) and Serious Adverse Events (SAE) graded using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE).
  The CTCAE has 5 grades with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1=Mild AE; Grade 2=Moderate AE; Grade 3=Severe AE; Grade 4=Life-threatening or disabling AE; and Grade 5=Death related to AE.
Time Frame: Subjects were followed for safety from enrollment for up to 8 months (9 three-week cycles plus 30 days after end of treatment)
Population: The total analysis population was 69 subjects: 70 subjects were enrolled; 45 were randomly assigned to treatment (24 to OGX-011/mitoxantrone and 21 to OGX-011 /docetaxel). An additional 25 subjects were assigned to OGX-011/docetaxel. One subject in the mitoxantrone arm was ineligible and did not receive study treatment.
Measure: Number; unit: percentage of participants
Groups:
- OGX-011 + Mitoxantrone + Prednisone: custirsen (OGX-011) in combination with mitoxantrone and prednisone
- OGX-011 + Docetaxel + Prednisone: custirsen (OGX-011) in combination with docetaxel and prednisone
Arm/Group | OGX-011 + Mitoxantrone + Prednisone | OGX-011 + Docetaxel + Prednisone
Number analyzed (Participants) | 23 | 46
percentage of participants
  Percent of Subjects with Serious Adverse Events | 26 | 26
  Percent of Subjects with Grade 5 Adverse Events | 13 | 4
  Percent of Subjects with Grade 4 Adverse Events | 26 | 15
  Percent of Subjects with Grade 3 Adverse Events | 70 | 52
  Percent of Subjects with Grade 2 Adverse Events | 83 | 98
  Percent of Subjects with Grade 1 Adverse Events | 100 | 100
  Percent of Subjects who Discontinued Study Drug | 22 | 17

2. Secondary Outcome: Feasibility of Treatment With Custirsen (OGX-011) in Combination With Second-line Chemotherapy Based on Prostate Specific Antigen (PSA) Response
Description: PSA or prostate specific antigen is a marker for prostate cancer. A PSA response was defined as a decrease in PSA values of ≥ 50% relative to baseline on two or more consecutive measurements that were 4-6 weeks apart.
Time Frame: PSA was evaluated at screening, on Day 1 of each cycle, at the end of treatment visit and during off-treatment follow up (up to 27 months)
Population: Subjects were evaluable for PSA response if they had baseline PSA and at least two post baseline PSA values.
  One subject was not evaluable for PSA response; he had only one post baseline PSA value. A PSA response was defined in the protocol as a decrease in PSA of ≥ 50% relative to baseline on two or more consecutive measurements 4-6 weeks apart.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OGX-011 / Mitoxantrone/Prednisone | OGX-011 / Docetaxel/Prednisone
Number analyzed (Participants) | 23 | 45
percentage of participants | 17 [5.0 to 38.8] | 31 [18.2 to 46.6]

3. Secondary Outcome: Feasibility of Treatment With OGX-011 in Combination With Either Docetaxel/Prednisone or Mitoxantrone/Prednisone as Second Line Chemotherapy Based on Time to Pain Progression
Description: Time to pain progression was defined as the time (months) from the first dose of OGX-011 to the first documentation of pain or analgesic progression or initiation of palliative radiation therapy. Pain response was defined as either a decrease of at least two points on the 11-point Worst Pain Scale, without an increase in analgesic level, maintained for at least two consecutive measurements approximately three weeks apart -or- a decrease in analgesic level, without an increase in pain score, maintained for at least two consecutive measurements approximately three weeks apart.
Time Frame: Enrollment until pain progression (up to 21 months)
Population: Subjects were evaluable for pain response if they had a baseline Worst Pain Score ≥ 2 or were on opioid analgesics at baseline.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | OGX-011 + Mitoxantrone + Prednisone | OGX-011 + Docetaxel + Prednisone
Number analyzed (Participants) | 18 | 20
months | 5.2 [1.6 to 8.1] | 7.2 [5.8 to 10.6]

4. Secondary Outcome: Relationship Between Changes in Serum Clusterin Levels and Change in Serum PSA Levels When OGX-011 in Combination With Either Docetaxel/Prednisone or Mitoxantrone/Prednisone is Administered as Second Line Chemotherapy.
Description: Serum clusterin samples were collected prior to receiving OGX-011 loading dose 1, prior to study treatment on Day 1 of each cycle, and at the end of treatment. PSA was evaluated at screening, on Day 1 of each cycle, at the end of treatment visit, and during off-treatment follow-up. PSA response was defined in the protocol as a decrease in PSA of ≥ 50% relative to baseline on two or more consecutive measurements 4-6 weeks apart.
Time Frame: Enrollment until disease progression (up to 13 months)
Population: All 69 subjects were included. Data are presented for the 20 subjects who achieved a 50% decline in PSA (6 subjects who received mitoxantrone and prednisone in combination with OGX-011 and 14 subjects who received docetaxel and prednisone in combination with OGX-011)
Measure: Number; unit: percentage of participants
Arm/Group | OGX-011 + Mitoxantrone + Prednisone | OGX-011 + Docetaxel + Prednisone
Number analyzed (Participants) | 23 | 46
percentage of participants
  Minimum clusterin level < or = to 45 mcg/mL | 22 | 24
  Minimum clusterin level > 45 mcg/mL | 4 | 7

ADVERSE EVENTS:
Arm/Group | OGX-011 / Mitoxantrone/Prednisone | OGX-011 / Docetaxel/Prednisone
Serious Adverse Events (participants affected / at risk) | 6/23 | 12/46
Other Adverse Events (participants affected / at risk) | 23/23 | 46/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OGX-011 / Mitoxantrone/Prednisone (N=23) | OGX-011 / Docetaxel/Prednisone (N=46)
Bronchiolitis (Infections and infestations) | 0 | 1
Klebsiella Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Acute Abdomen (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 1
Death (General disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OGX-011 / Mitoxantrone/Prednisone (N=23) | OGX-011 / Docetaxel/Prednisone (N=46)
Fatigue (General disorders) | 18 | 32
Oedema Peripheral (General disorders) | 10 | 21
Chills (General disorders) | 10 | 19
Pyrexia (General disorders) | 14 | 14
Asthenia (General disorders) | 3 | 7
Chest Pain (General disorders) | 3 | 0
Mucosal Inflammation (General disorders) | 3 | 0
Pain (General disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 14 | 23
Vomiting (Gastrointestinal disorders) | 10 | 16
Diarrhoea (Gastrointestinal disorders) | 5 | 19
Constipation (Gastrointestinal disorders) | 4 | 10
Abdominal Pain (Gastrointestinal disorders) | 6 | 3
Stomatitis (Gastrointestinal disorders) | 2 | 4
Abdominal Distension (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Bone Pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Neuropathy Peripheral (Nervous system disorders) | 3 | 13
Dysgeusia (Nervous system disorders) | 3 | 12
Dizziness (Nervous system disorders) | 3 | 11
Headache (Nervous system disorders) | 7 | 4
Hypoaesthesia (Nervous system disorders) | 2 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 2 | 0
Neuralgia (Nervous system disorders) | 0 | 3
Syncope (Nervous system disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 12 | 16
Dehydration (Metabolism and nutrition disorders) | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 9
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Oral Herpes (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 2 | 2
Weight Decreased (Investigations) | 6 | 8
Aspartate Aminotransferase Increased (Investigations) | 2 | 0
Insomnia (Psychiatric disorders) | 8 | 5
Anxiety (Psychiatric disorders) | 4 | 6
Depression (Psychiatric disorders) | 2 | 4
Confused State (Psychiatric disorders) | 2 | 1
Mood Altered (Psychiatric disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 8 | 8
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Hypotension (Vascular disorders) | 1 | 5
Hot Flush (Vascular disorders) | 4 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 6
Fall (Injury, poisoning and procedural complications) | 0 | 3
Lacrimation Increased (Eye disorders) | 1 | 8
Haematuria (Renal and urinary disorders) | 1 | 3
Pollakiuria (Renal and urinary disorders) | 2 | 1
Nocturia (Renal and urinary disorders) | 2 | 0
Pelvic Pain (Reproductive system and breast disorders) | 2 | 2
Atrial Fibrillation (Cardiac disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All investigators had an agreement with the Canadian Urological Oncology Group (CUOG). The investigators were to provide CUOG with text to be presented or published 45 days prior to the release for review. Results from one institution were not to be presented before the multi-center publication. If there is no multi-center publication within 12 months after the Study completion the Investigator had the right to publish the results.